CLINICAL TRIAL: NCT01961726
Title: A Phase I/II Study to Evaluate the Safety and Efficacy of JVS-100 Administered by Retrograde Delivery to Cohorts of Adults With Ischemic Heart Failure
Brief Title: Study to Evaluate the Safety and Efficacy of JVS-100 Administered to Adults With Ischemic Heart Failure
Acronym: RETRO-HF
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Juventas Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JTCS-003
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Ischemic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Biological: 30 mg dose of JVS-100; Biological: 45 mg dose of JVS-100
- 30 mg dose of JVS-100 (Experimental)
  Interventions: Biological: Placebo; Biological: 45 mg dose of JVS-100
- 45 mg dose of JVS-100 (Experimental)
  Interventions: Biological: Placebo; Biological: 30 mg dose of JVS-100

INTERVENTIONS:
Biological: Placebo — Coronary Sinus Delivery
  Arms: 30 mg dose of JVS-100; 45 mg dose of JVS-100
Biological: 30 mg dose of JVS-100 — Coronary Sinus Delivery
  Arms: 45 mg dose of JVS-100; Placebo
Biological: 45 mg dose of JVS-100 — Coronary Sinus Delivery
  Arms: 30 mg dose of JVS-100; Placebo

SUMMARY:
A phase I/II study to evaluate the safety and efficacy of JVS-100 administered by retrograde delivery to cohorts of adults with Ischemic Heart Failure.

DETAILED DESCRIPTION:
72 subjects with ischemic cardiomyopathy. The Phase I portion (n=12 subjects) will be open label. In the first cohort, six subjects will receive a single dose of 30 mg of JVS-100 with a minimum of 3 days between each enrollment. After seven days following the enrollment of the last patient of cohort 1, a safety assessment by the DSMC will be performed. Upon DSMC approval, the second cohort of six subjects will receive a single dose of 45 mg of JVS-100 with a minimum of 3 days between each enrollment. After seven days following the enrollment of the last patient of cohort 2, a safety assessment by the DSMC will be performed. Upon DSMC approval, up to 60 subjects will be randomized (1:1:1) to receive a single dose of 30 mg or 45 mg of JVS-100 or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign informed consent
* Greater than or equal to 18 years of age
* Poor quality of life as measured by the Minnesota Living with Heart Failure Questionnaire (MLWHFQ)
* Impaired 6 Minute Walk test
* Ischemic cardiomyopathy without an acute coronary syndrome within the last 6 months
* Residual well-demarcated region of LV systolic dysfunction defined as at least 3 consecutive segments of abnormal wall motion by echocardiography read at the echocardiography core laboratory
* LVEF less than or equal to 40% measured by echocardiography read at the echocardiography core laboratory
* Subject receiving stable optimal pharmacological therapy defined as:

  * ACE inhibitor and/or ARB, and Beta-blocker for 90 days with stable dose* for
  * 30 days unless contraindicated
  * Diuretic in subjects with evidence of fluid retention
  * ASA unless contraindicated
  * Statin unless contraindicated
  * Aldosterone antagonist per physician discretion
* Subject must not have a permanent device placed in the coronary sinus at the time of enrollment *As defined as no more than 50% change in dose

Exclusion Criteria:

* Planned revascularization within 30 days following enrollment

  * Note: if an angiographic study has been performed within the last year and the subject is enrolled, the angiography study report should be included as part of the subject's file
* Estimated Glomerular Filtration Rate < 30 ml/min*
* Signs of acute heart failure within 24 hours of scheduled infusion
* History of aortic valve regurgitation classified as "moderate-severe" or worse
* Patients will be excluded who have:

  * Known prior trauma to the coronary sinus
  * In dwelling instrumentation that may hamper coronary venous catheterization, including a biventricular pacing coronary sinus lead
* Mitral regurgitation defined as "severe" measured by echocardiography at the clinical site
* Patients with planned mitral valve repair or replacement surgery
* Any patient with a history of cancer will be excluded unless:

  * The cancer was limited to curable non-melanoma skin malignancies and/or
  * The cancer was removed by a successful tumor resection, with or without radiation or chemotherapy treatment, 5 years or more prior to enrollment in this study without recurrence.
* Subjects with persistent (per ACC/AHA/EEC guidelines)53, defined as recurrent AF episodes lasting longer than 7 days) or chronic atrial fibrillation will be excluded unless:

  * A stable, regular heart rate is maintained with a biventricular pacemaker
  * A stable, regular heart rate is maintained with a univentricular pacemaker pacing less than or equal to 40% of the time
* Inability to undergo 6 minute walk or treadmill exercise test
* Previous solid organ transplant
* Subjects with greater than 40% univentricular RV Pacing
* Subjects with uncontrolled diabetes defined as HbA1c >10 %
* Participation in an experimental clinical trial within 30 days prior to enrollment
* Life expectancy of less than 1 year
* Positive pregnancy test (serum βHCG) in women of childbearing potential and/or unwillingness to use contraceptives or limit sexual activity as described in Section 8.2.1 below
* Unwillingness of men capable of fathering a child to agree to use barrier contraception or limit sexual activity as described in Section 8.2.1 below
* Subjects who are breast feeding
* Subjects with a positive test results for hepatitis B/C and/or HIV will be excluded unless:

  * The subject is a carrier for hepatitis B/C but has never had an active flare
* Subjects with a history of Systemic Lupus Erythematosus (SLE) flare
* Total Serum Bilirubin >4.0 mg/dl
* Aspartate aminotransferase (AST) > 120 IU/L
* Alanine aminotransferase (ALT) > 135 IU/L
* Alkaline phosphatase (ALP): >300 IU/L
* Clinically significant elevations in PT or PTT relative to laboratory norms at day 0
* Critical limb ischemia that limits the patients from completing 6 minute walk or treadmill testing
* Subjects with severe chronic obstructive pulmonary disease (COPD)

  * Severe defined as having been hospitalized for COPD within the last 12 months
* Any subject requiring home oxygen use for treatment of the symptoms of COPD
* History of drug or alcohol abuse within the last year
* A subject will be excluded if he/she is unfit for the trial based on the discretion of the site Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Impact of JVS-100 delivery on 6 minute walk distance at 4 month follow-up | 4 Months
  To investigate the impact of single doses of JVS-100 (either 30 or 45 mg) delivered retrograde via the coronary sinus through the Oscor Venos Occlusion Balloon catheter on 6 minute walk distance compared to placebo at 4 months post dosing.

SECONDARY OUTCOMES:
Impact of JVS-100 delivery on heart failure symptoms compared to placebo at 4 and/or 12 month follow-up | 4 and/or 12 months
  To assess the impact of a single dose of JVS-100 on heart failure symptoms compared to placebo at 4 and/or 12 months post-dosing.

OTHER OUTCOMES:
Impact of JVS-100 delivery on quality of life measure at 4 month follow-up | 4 Months
  To investigate the impact of single doses of JVS-100 (either 30 or 45 mg) delivered retrograde via the coronary sinus through the Oscor Venos Occlusion Balloon catheter on quality of life measure compared to placebo at 4 months post dosing.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Cardiology, P.C., Birmingham, Alabama
  - University of Florida, Gainsville, Florida
  - The Carl and Edyth Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah